CLINICAL TRIAL: NCT02030275
Title: A Multi-Center, Prospective, Randomized, Double-Blind, Within-Subject Controlled, Phase 2a Study to Evaluate the Effectiveness and Safety of RXI 109 on the Outcome of Scar Revision Surgery on Transverse Hypertrophic Scars on the Lower Abdomen Resulting From Previous Surgeries in Healthy Adults
Brief Title: A Study to Evaluate the Effectiveness and Safety of RXI 109 on the Outcome of Scar Revision Surgery in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RXi Pharmaceuticals, Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RXI-109-1301
Record Dates: First submitted 2014-01-06; First posted 2014-01-08 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Hypertrophic Scar
Keywords: Hypertrophic scar; Cicatrix; Scar prevention; Scar revision
MeSH Terms: conditions — Cicatrix, Hypertrophic; Cicatrix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RXI-109 (Experimental): Treatment with RXI-109 on one side of revised scar and a placebo comparator on the other side. Treatment to begin either immediately or 2 weeks following the scar revision surgery.
  Interventions: Drug: RXI-109
- Placebo (Placebo Comparator): Treatment with RXI-109 on one side of revised scar and a placebo comparator on the other side. Treatment to begin either immediately or 2 weeks following the scar revision surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RXI-109 — surgery.
  Arms: RXI-109
Drug: Placebo — surgery.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effectiveness of RXI-109 in reducing the recurrence of hypertrophic scar formation following elective revision of a pre-existing hypertrophic abdominal scar.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 21-55 years of age in general good health
* Previous partial hysterectomy, Cesarean section or abdominoplasty surgery resulting in a transverse hypertrophic scar of ≥ 11 cm in length
* Scar to be revised must have been present for > 9 months

Exclusion Criteria:

* Use of tobacco or nicotine-containing products
* Pregnant or lactating
* Post-menopausal or full hysterectomy

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2013-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Reduction in recurrence of hypertrophic scarring after scar revision surgery | 9 months
  To evaluate the effectiveness of RXI-109 in reducing the recurrence of hypertrophic scar formation following elective revision of a hypertrophic abdominal scar

SECONDARY OUTCOMES:
Safety of RXI-109 | 9 months
  To assess severity and frequency of reported adverse events and clinically-relevant changes in laboratory testing after elective revision of a hypertrophic abdominal scar

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Pavco, PhD, Study Director — RXi Pharmaceuticals
Locations (5):
- United States (4):
  - Lake Worth, Florida
  - Chicago, Illinois
  - St Louis, Missouri
  - Huntersville, North Carolina
- San Pedro Sula, Honduras